CLINICAL TRIAL: NCT04038996
Title: A Single-Center, Prospective, Observational Trial to Analyze the Relationship Between Single Nucleotide Polymorphism rs2910164 and the Efficacy and Safety of Immune Checkpoint Inhibitor Therapy
Brief Title: The Role of SNP rs2910164 in Patients Treated With Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Head of Department of Tumorimunnology and Immunoregulation, University of Freiburg
Other Study IDs: SNP_irAE
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cancer
Keywords: immune checkpoint inhibitor; single nucleotide polymorphism; microRNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The rs2910164 genotype will be assessed using DNA isolated from peripheral blood samples and Taqman realtime PCR assays.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to investigate whether the SNP rs2910164 in the pre-miR-146a gene is associated with outcome and toxicity of immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
The single nucleotide polymorphism (SNP) rs2910164 within the gene for microRNA-146a (miR-146a) reduces miR-146a expression. Previous studies of the investigators demonstrated that this SNP was associated with increased acute GvHD severity in patients undergoing allogeneic hematopoietic stem cell transplantation. In this prospective, observational study the investigators aim to analyze, whether SNP rs2910164 is associated with severity of immune-related adverse events of immune checkpoint inhibitor therapy. Moreover, association of rs2910164 with outcome parameters will be studied.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of cancer
* treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PD-L1 or anti-CTLA4)
* age ≥ 18 years
* peripheral blood sample available
* written informed consent
* ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* lack of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer undergoing immune checkpoint inhibitor therapy
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Severity of immune-related adverse events (irAEs) | 2 years
  according to CTCAE
Progression-free survival (PFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, MD, Principal Investigator — University of Freiburg

REFERENCES:
- [Background] Jazdzewski K, Murray EL, Franssila K, Jarzab B, Schoenberg DR, de la Chapelle A. Common SNP in pre-miR-146a decreases mature miR expression and predisposes to papillary thyroid carcinoma. Proc Natl Acad Sci U S A. 2008 May 20;105(20):7269-74. doi: 10.1073/pnas.0802682105. Epub 2008 May 12. PMID 18474871
- [Background] Stickel N, Hanke K, Marschner D, Prinz G, Kohler M, Melchinger W, Pfeifer D, Schmitt-Graeff A, Brummer T, Heine A, Brossart P, Wolf D, von Bubnoff N, Finke J, Duyster J, Ferrara J, Salzer U, Zeiser R. MicroRNA-146a reduces MHC-II expression via targeting JAK/STAT signaling in dendritic cells after stem cell transplantation. Leukemia. 2017 Dec;31(12):2732-2741. doi: 10.1038/leu.2017.137. Epub 2017 May 9. PMID 28484267
- [Result] Marschner D, Falk M, Javorniczky NR, Hanke-Muller K, Rawluk J, Schmitt-Graeff A, Simonetta F, Haring E, Dicks S, Ku M, Duquesne S, Aumann K, Rafei-Shamsabadi D, Meiss F, Marschner P, Boerries M, Negrin RS, Duyster J, Zeiser R, Kohler N. MicroRNA-146a regulates immune-related adverse events caused by immune checkpoint inhibitors. JCI Insight. 2020 Mar 26;5(6):e132334. doi: 10.1172/jci.insight.132334. PMID 32125286